CLINICAL TRIAL: NCT03556813
Title: Artificial Intelligence vs Physicians for Breast Cancer Patients' Information : a Blind, Randomized, Controlled Study
Brief Title: Artificial Intelligence vs Physicians for Breast Cancer Patients' Information
Status: Completed | Type: Observational
Sponsor: Wefight (Industry)
Responsible Party: Sponsor
Other Study IDs: INCASE0518
Record Dates: First submitted 2018-05-31; First posted 2018-06-14 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
Keywords: Patient information; Natural Language Processing; Conversational agent; Chatbot
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group Vik: women over the age of 18 with breast cancer or remission
  Interventions: Other: survey
- Group physicians: women over the age of 18 with breast cancer or remission
  Interventions: Other: survey

INTERVENTIONS:
Other: survey — non-inferiority study, randomized, blind, excluding health product, with no risk or constraint, in which all the acts are performed in the usual way and do not modify the patient's management.

SUMMARY:
Chatbots (contraction of "chat" and "robot") are a computer software program that use statistical learning and aim to simulate a conversation by text or voice message. The use of these chatbots was evaluated as part of the increase in therapeutic adherence and information on well-being and mental health.

In clinical studies, chatbots are useful in gathering information through questionnaires directly submitted during conversations or through keyword analyzes. There is no longer any delay between the moment the patient notices a side effect, for example, and the moment when the patient announces it during a consultation. The responses given by the chatbot do not constitute medical advice and only provide information on the treatments envisaged or in progress in the context of the management of breast cancer.

The main objective of the study is to show that the chatbot Vik's answers to the common questions asked by breast cancer patients about their therapeutic management are at least as satisfactory as answers given by a committee of multidisciplinary doctors

DETAILED DESCRIPTION:
A total of 20 most frequently asked questions will be defined on a cohort of 150 breast cancer patients. These questions will be asked on the one hand to the chatbot Vik and on the other hand to a multidisciplinary medical committee (surgeon oncologist, medical oncologist and oncologist radiotherapist). The scientific quality of the responses of the two groups will be validated by a second multidisciplinary group of physicians, independent of the first.

A cohort of 150 patients will then be randomized blind and in 1 to 1 to receive the responses of the chatbot Vik and the answers of the doctors' committee. Each patient will then have to answer the EORTC QLQ-INFO255-7 questionnaire, evaluating the quality of the medical information.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years
* paitents with breast cancer

Exclusion Criteria:

* Patient unable to formulate his opposition
* Patient with cancer other than breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with breast cancer or in remission
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-01-20 (Actual)

PRIMARY OUTCOMES:
Quality of Patient information | Through study completion, an average of 3 months
  The quality of the participating patient's information about their disease and their treatment will be assessed using the standardized EORTC QLQ-INFO25 survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Wefight, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bibault JE, Chaix B, Guillemasse A, Cousin S, Escande A, Perrin M, Pienkowski A, Delamon G, Nectoux P, Brouard B. A Chatbot Versus Physicians to Provide Information for Patients With Breast Cancer: Blind, Randomized Controlled Noninferiority Trial. J Med Internet Res. 2019 Nov 27;21(11):e15787. doi: 10.2196/15787. PMID 31774408